CLINICAL TRIAL: NCT03797911
Title: Efficacy of Resistive Capacitive Monopolar Radiofrequency in the Physiotherapeutic Treatment of Chronic Pelvic Pain: Randomized Clinical Trial.
Brief Title: Efficacy of Resistive Capacitive Monopolar Radiofrequency in the Physiotherapeutic Treatment of Chronic Pelvic Pain: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAPbarcelona (Other)
Responsible Party: Principal Investigator, Andrea Carralero Martínez, Physical therapist, RAPbarcelona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAP39426977
Record Dates: First submitted 2018-12-12; First posted 2019-01-09 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Pelvic Pain; Pelvic Pain Syndrome; Chronic Pain; Chronic Pain Syndrome; Chronic Pelvic Inflammatory Disease; Physical Therapy
MeSH Terms: conditions — Pelvic Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active resistive capacitive monopolar radiofrequency (Experimental): Application of the technique in the intervention group (activated resistive capacitive monopolar radiofrequency therapy): The intervention group will receive the treatment with activated resistive capacitive monopolar radiofrequency system, with the resistive electrode at the minimum intensity, together with the techniques of conventional physiotherapy treatment (trigger point treatment and myofascial techniques according to the location of pain) and pain education.
  The patient will be stretched on the stretcher and the session will last 45 minutes, once a week, for 10 sessions. Ass baseline, after half therapy and after 10 weeks therapy.
  Interventions: Combination Product: Active resistive capacitive monopolar radiofrequency with physiotherapeutic techniques and pain education
- Inactive resistive capacitive monopolar radiofrequency (Placebo Comparator): Application of the technique in the control group (inactivated resistive capacitive monopolar radiofrequency therapy): The control group will receive the treatment with inactivated resistive capacitive monopolar radiofrequency system (placebo), with the resistive electrode at the minimum intensity, together with the techniques of conventional physiotherapy treatment (trigger point treatment and myofascial techniques according to the location of pain) and pain education.
  The patient will be stretched on the stretcher and the session will last 45 minutes, once a week, for 10 sessions. Ass baseline, after half therapy and after 10 weeks therapy.
  Interventions: Combination Product: Inactive resistive capacitive monopolar radiofrequency with physiotherapeutic techniques and pain education

INTERVENTIONS:
Combination Product: Active resistive capacitive monopolar radiofrequency with physiotherapeutic techniques and pain education — Activated resistive capacitive monopolar radiofrequency is applied to the patient along with the conventional treatment of physiotherapeutic techniques and pain education.
  Arms: active resistive capacitive monopolar radiofrequency
Combination Product: Inactive resistive capacitive monopolar radiofrequency with physiotherapeutic techniques and pain education — Disactivated resistive capacitive monopolar radiofrequency inactived is applied to the patient along with the conventional treatment of physiotherapeutic techniques and pain education.
  Arms: Inactive resistive capacitive monopolar radiofrequency

SUMMARY:
This study evaluates if the application of resistive capacitive monopolar radiofrequency therapy associated with physiotherapeutic techniques and pain education provides benefits with respect to physiotherapy and pain education techniques alone in the management of patients with chronic pelvic pain.

DETAILED DESCRIPTION:
It is evident that physiotherapeutic techniques and pain education are a first-line treatment for patients suffering from chronic pelvic pain. But there is no scientific evidence that resistive capacitive monopolar radiofrequency can be another treatment option for these patients, although at the clinical level there is evidence of its beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

* Have an age equal to or greater than 18 years
* Having chronic pelvic pain of six or more months of evolution.

Exclusion Criteria:

* Failure to grant informed consent.
* Have fibromyalgia.
* Present a pacemaker or other type of electronic implant.
* Suffer systemic diseases (infectious, vascular, endocrine, metabolic or neoplastic conditions).
* Previous treatment with chemotherapy and / or radiotherapy in the pelvic area.
* Suffering from neuromuscular diseases (amyotrophic lateral sclerosis, multiple sclerosis, myasthenia gravis or spinal muscular atrophy).
* Have myelopathy and osteomyelitis.
* Have neurological and / or metabolic pathology that alters the response capacity: diabetes, parkinson's disease, senile dementia ...
* Have an alteration of the central nervous system (traumatic or spinal vascular injury)
* Suffer oncological processes with sacral involvement.
* Have a severe mental disorder.
* Have vulvodynia
* Be pregnant.
* Have undergone surgery in the last 3 months in the pelvic area.
* Have hypersensitivity of the skin, hyposensitivity and / or rejection of manual contact.
* Inability to correctly complete the questionnaires or understand the study protocol.
* Having initiated other pelvic physiotherapy treatments during the study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-03-23 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Efficacy of resistive capacitive monopolar radiofrequency in the modification of the perception of pain | baseline and 10 weeks
  The objective is to assess if there is a change in the perception of pain intensity according to VAS (Visual Analog Scale). Compare baseline and at the end of the intervention.
  The Visual Analog Scale is a validated questionnaire that scores between 0 and 10 the perception of pain that the patient has. In a line of 10 cm the patient will mark his intensity of the pain taking into account that 0 means "I have no pain" and 10 means "I have an unbearable pain".
  The Visual Analog Scale (VAS) suitably collects the pain intensity perceived by the patient and allows to assess the severity of the disease, as well as the improvement obtained with the treatment.

SECONDARY OUTCOMES:
Assess quality of life | baseline, 5 and 10 weeks
  Asess the perceived quality of life of patients in the study according to the SF-12 questionnaire.
  The Short-Form 12 Health Survey was designed in 1994 with the aim that, through the self-completion of a brief questionnaire, the perception of physical and mental quality of life could be objectified in a simpler way than the original questionnaire SF -36. This simple questionnaire of 12 items representing the 8 dimensions of health was originally developed in English. It is a questionnaire that has proven to be valid and reliable to be used in clinical practice as an instrument to assess the quality of life. The 8 dimensions are the physical function (2 items), physical role (2 items), body pain (1 item), general health (1 item), vitality (1 item), social function (1 item), emotional role (2) items) and mental health (2 items). The result is two variables (physical and mental) that value quality in these two aspects.
Assess kinesiophobia | baseline, 5 and 10 weeks
  Asess the kinesiophobia suffered by patients in the study according to the TSK-11 (Tampa Scale of Kinesiophobia) questionnaire.
  The Tampa Scale of Kinesiophobia (TSK-11), validated in Spanish, adequately captures the patient's movement capacity taking into account the perceived pain intensity in 11 questions. It is a tool that allows assessing the severity of the disease, as well as the improvement that is obtained with the treatment.
Assess catastrophism | baseline, 5 and 10 weeks
  Asess the catastrophism suffered by patients in the study according to the Catastrophism scale.
  The Catastrophism Scale, also validated in Spanish, allows us to assess the catastrophic intensity of the disease, a more psychological aspect, but also very relevant in this chronic and disabling pathology. It is a tool that allows assessing the severity of the disease, as well as the improvement that is obtained with the treatment. It is a questionnaire of 20 questions.
Assess the degree of adherence to treatment | 10 weeks
  Assess the degree of adherence to treatment (%) of the patients who are in this study.
Assess number of participants with high adherence to treatment | 10 weeks
  Assess the number of patients (n) with high adherence who are in this study.
Assess number of participants with adverse effects | 10 weeks
  Evaluate and identify the number of participants (n) who have an adverse effect during the study intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Andrea Carralero Martinez, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carralero-Martinez A, Naranjo-Ortiz C, Blanco-Ratto L, Kauffmann S, Ramirez-Garcia I. Assessing Kinesiophobia and Catastrophizing Patient-Reported Outcomes in a Randomized Controlled Trial: Efficacy of Capacitive-Resistive Monopolar Radiofrequency Combined with Myofascial Techniques vs. Sham Radiofrequency in Chronic Pelvic Pain Syndrome-A Secondary Analysis. Int Urogynecol J. 2025 Apr;36(4):799-811. doi: 10.1007/s00192-025-06052-x. Epub 2025 Jan 28. PMID 39873778
- [Derived] Carralero-Martinez A, Munoz Perez MA, Pane-Alemany R, Blanco-Ratto L, Kauffmann S, Ramirez-Garcia I. Efficacy of capacitive resistive monopolar radiofrequency in the physiotherapeutic treatment of chronic pelvic pain syndrome: study protocol for a randomized controlled trial. Trials. 2021 May 20;22(1):356. doi: 10.1186/s13063-021-05321-6. PMID 34016168